CLINICAL TRIAL: NCT04132427
Title: Microbiota Transfer Therapy for Children With Both Pitt Hopkins Syndrome and Gastrointestinal Disorders
Brief Title: MTT for Children With Both Pitt Hopkins Syndrome and Gastrointestinal Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Pitt Hopkins Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#: 120190263
Record Dates: First submitted 2019-10-11; First posted 2019-10-18 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-03

CONDITIONS: Pitt Hopkins Syndrome
Keywords: microbiota transfer therapy; fecal transplant; fecal microbiota transplant; intestinal microbiota
MeSH Terms: conditions — Pitt-Hopkins syndrome | interventions — Vancomycin; magnesium citrate; Microbiota

STUDY DESIGN:
Intervention Model Description: Part 1: Randomized, double-blind, placebo-controlled Part 2: Treatment group enters observation, placebo group switched to treatment Part 3: Long-term observation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is double-blind Parts 2 and 3 are single-blind (outcomes assessor is blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Treatment (Experimental): Vancomycin, magnesium citrate, microbiota
  Interventions: Combination Product: vancomycin, magnesium citrate, microbiota
- Group B: Placebo (Placebo Comparator): placebo vancomycin, real magnesium citrate (because it obviously empties the bowels) and placebo microbiota
  Interventions: Combination Product: placebo vancomycin, real magnesium citrate, placebo microbiota

INTERVENTIONS:
Combination Product: vancomycin, magnesium citrate, microbiota — 10 days of oral vancomycin, then 1 day of oral magnesium citrate, , then 4 days of high-dose oral microbiota, followed by 12 weeks of low-dose oral microbiota
  Arms: Group A: Treatment
Combination Product: placebo vancomycin, real magnesium citrate, placebo microbiota — 10 days of oral placebo vancomycin, then 1 day of oral real magnesium citrate, , then 4 days of high-dose oral placebo microbiota, followed by 12 weeks of low-dose oral placebo microbiota
  Arms: Group B: Placebo

SUMMARY:
The investigators propose to investigate Microbiota Transfer Therapy (MTT) for treating patients with Pitt Hopkins Syndrome (PTHS) and gastrointestinal problems similar to Irritable Bowel Syndrome (IBS). MTT involves a combination of 10 days of oral vancomycin (an antibiotic to kill pathogenic bacteria), followed by a bowel cleanse, followed by 12 weeks of Fecal Microbiota (FM).

DETAILED DESCRIPTION:
For children ages 5-17 years with PTHS and gastrointestinal problems, a Phase 2 clinical trial will evaluate the safety, tolerability, and efficacy of MTT.

Randomized, double-blind, placebo-Controlled Treatment (14 weeks)

The trial will be a randomized, double-blind, placebo-controlled trial which will include a 10-day treatment with oral vancomycin (or placebo), then 1 day of magnesium citrate to cleanse the bowel of vancomycin and bacteria/feces (all participants, since its bowel-emptying effect cannot be blinded), followed by oral administration of FM (or placebo). An initial high dose of FM (or placebo) for two days will be followed by a lower maintenance dose of FM (or placebo) for 12 weeks.

Group A: real treatment Group B: placebo vancomycin, real magnesium citrate, placebo FM

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 7-17 years with Pitt Hopkins Syndrome (verified by genetic testing)
2. GI disorder as defined below that has lasted for at least 2 years.
3. No changes in medications, supplements, diet, or therapies in last 2 months, and no intention to change them during the Parts 1 and 2 of the clinical trial.
4. Ability to swallow pills (without chewing)
5. Review of last two years of medical records by the study physician.

Exclusion Criteria:

1. Antibiotics in last 3 months
2. Probiotics in last 2 months, or fecal transplant in last 12 months
3. Tube feeding
4. Severe gastrointestinal problems that require immediate treatment (life-threatening)
5. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions
6. Unstable, poor health (based on study physician's opinion)
7. Recent or scheduled surgeries
8. Current participation in other clinical trials
9. Females who are pregnant or who are at risk of pregnancy and sexually active without effective birth control.
10. Allergy or intolerance to vancomycin or magnesium citrate
11. Clinically significant abnormalities at baseline on two blood safety tests: Comprehensive Metabolic Panel, and Complete Blood Count with Differential.
12. Evidence of significant impairment of immune system, or taking medications that can compromise the immune system, and thus increase risk if exposed to multiple-drug resistant bacteria.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: link for our research group — https://autism.asu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: Treatment | Group B: Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Treatment | Group B: Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (3.6) | 12.7 (3.1) | 12.8 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Daily Stool Record [Mean (Standard Deviation); unit: Number of abnormal days out of 14 days] | 14 (0) | 14 (0) | 14 (0)

OUTCOME MEASURES:

1. Primary Outcome: Daily Stool Record (DSR(
Description: The DSR is a daily record of their bowel movements including Bristol Stool Form scale. It is rated as the number of days (out of 14 days) with an abnormal report (abnormal stool, no stool, or the use of a gastrointestinal treatment). A higher percentage indicates worse symptoms.
Time Frame: change in % abnormal days from baseline (for 2 weeks) vs. week 14 (2 weeks from week 13-14)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
days | -2.3 (2.5) | 0 (0)

2. Primary Outcome: Safety Measures
Description: number of adverse events and serious adverse events likely associated with treatment
Time Frame: weeks 0-14
Measure: Number; unit: number of AEs among all participants
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
number of AEs among all participants | 8 | 10

3. Secondary Outcome: CGI for GI Disorders
Description: Clinical Global Impressions of GI Disorders, including severity, change in severity, and side effects. The severity is rated on a scale of 1-7, with 1 being normal and 7 being the worst possible.
Time Frame: change in score between baseline and week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | -1 (1) | -.67 (1.15)

4. Secondary Outcome: CGI for PTHS Symptoms
Description: Clinical Global Impressions of Pitt Hopkins Syndrome symptoms, including severity, change in severity, and side effects. The severity is rated on a scale of 1-7, with 1 being normal and 7 being the worst possible.
Time Frame: change in score between baseline and week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 0 (0) | -.33 (.58)

5. Secondary Outcome: PGI-PTHS
Description: Parent Global Impressions of Pitt Hopkins Syndrome symptoms. This is a rating of 29 symptoms, and an average is computed. The scale ranges from -3 (much worse) to +3 (much better).
Time Frame: change in score between baseline and week 14
Measure: Mean (Standard Deviation); unit: -3 to +3
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
-3 to +3 | .68 (.97) | .29 (.44)

6. Secondary Outcome: GSRS
Description: Gastrointestinal Symptom Rating Scale. This is a 15-item questionnaire, with each item rated on a scale of 1 (no symptoms) to 7 (very severe discomfort). The average score for all 15 items is reported here.
Time Frame: change in score between baseline and week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | -2.3 (.87) | -1.07 (1.91)

7. Secondary Outcome: FLACC
Description: Revised Face Legs Activity Crying Consolability Pain Questionnaire for Children with Cognitive Impairment (FLACC). This is a rating scale of 5 symptoms of pain, with each item rated on a scale of 0 (no symptom) to 2 (maximum symptom), and the scores for each item are summed to create a total score (zero to 10).
Time Frame: change in score between baseline and week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Treatment | Group B: Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | -4.0 (2.65) | -2.67 (2.08)

ADVERSE EVENTS:
Time Frame: AE data reported here is from the start of the treatment to the end of treatment (approximately 14 weeks).
Description: We use standard definition of the Adverse events and Serious Adverse events.
Arm/Group | Group A: Treatment | Group B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Treatment (N=3) | Group B: Placebo (N=3)
Hyperactivity (Psychiatric disorders) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2)
Gassy (Gastrointestinal disorders) | 2 (2) | 2 (2)
Insomnia (General disorders) | 1 (1) | 2 (2)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Redness- Genitalia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Change in Stool Color (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04132427/Prot_SAP_000.pdf